CLINICAL TRIAL: NCT03093675
Title: Robotic Assisted Surgery for Treatment of Gynecological Diseases: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TELELAP-ALF-X
Record Dates: First submitted 2017-03-16; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Adnexal Diseases; Uterine Diseases
MeSH Terms: conditions — Adnexal Diseases; Uterine Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TELELAP ALF-X Robotic Surgical System (Experimental): The patients will undergo surgical procedures using the innovative TELELAP ALF-X robotic system.
  Interventions: Device: TELELAP ALF-X Robotic Surgical System

INTERVENTIONS:
Device: TELELAP ALF-X Robotic Surgical System — The surgical procedures will be performed using the innovative TELELAP ALF-X robotic system, equipped with multiple independent arms. Initial entry will be through a classic open in which the arm with the video camera will be inserted. The device has four independent arms (one for the video camera and three for surgical instruments). Patients will be in the lithotomy position, supported by Allen stirrups and under general anesthesia. The uterus will be manipulated with a multi-use uterine manipulator. After having induced a pneumoperitoneum, high-definition 3D-technology optics will be inserted. Three laparoscopic instruments will be used to complete the procedure. Standard techniques will be used.

SUMMARY:
This is a prospective, single-center clinical trial. One hundred and fifty patients affected by adnexal and uterine diseases will be recruited to undergo treatment with robotic assisted laparoscopic procedures using the innovative TELELAP ALF-X Endoscopic Robotic Surgical System with the primary objective of assessing the feasibility, efficacy and safety of this approach.

DETAILED DESCRIPTION:
The study proposed comprises a prospective, single-center clinical trial (Catholic University of the Sacred Heart of Rome, A. Gemelli University Polyclinic).

One hundred and fifty patients affected by adnexal and uterine diseases will be recruited to undergo treatment with robotic assisted laparoscopic procedures using the innovative TELELAP ALF-X Endoscopic Robotic Surgical System with the primary objective of assessing the feasibility, efficacy and safety of this approach.

Post-operative pain will be reported by the patients through a Visual Analog Scale (VAS). It will be assessed at 2, 4 and 12 and 24 hours after the procedure.

At the end of patient recruitment, surgical procedure times, the technical limits encountered, estimated blood loss, intra- and post-operative complications and the percentage of conversions from the standard laparoscopic approach to multiple access and/or to a laparotomic approach will be analyzed in order to arrive at the feasibility and efficacy of robotic assisted treatment.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age ≥ 18 years old
* Sign the informed consent form
* BMI ≤ 40
* A.S.A. Class < III or IV

Disease Inclusion Criteria:

* Ovarian cyst (enucleation/oophorectomy)
* Prophylactic bilateral oophorectomy
* Ectopic pregnancy (salpingotomy/salpingectomy)
* Tubal inflammatory disease (salpingotomy/salpingectomy)
* Infertility and sterility (treatment of endometriosis, chromo-salpingography, etc.)
* Benign uterine disease (Fibromatosis, Adenomyosis)
* Endometrial hyperplasia
* Stage Ia G1-2 Endometrial tumors
* Precancerous lesions of the uterine cervix
* Stage Ia uterine cervical tumors
* Pelvic endometriosis

Patient Exclusion Criteria:

* Pregnancy
* Liver disease
* Coagulation disorders
* Patient internal or anatomical criteria that preclude a laparoscopic approach

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study concerns female-only diseases, adnexal and uterine diseases
Enrollment: 150 (Actual)
Dates: Start 2013-10-23 (Actual); Primary Completion 2014-12-09 (Actual); Study Completion 2014-12-09 (Actual)

PRIMARY OUTCOMES:
Feasibility and complications of robotic assisted surgery in the treatment of gynecological diseases | Pre-operative to 30 days follow-up
  The rate of complications and conversions to laparoscopic/laparotomic surgery will be collected and calculated. As this is a pilot study, no pre-determined success criteria has been set. The number of complications observed during robotic assisted surgery in the treatment of gynecological diseases will be registered.

SECONDARY OUTCOMES:
Robotic assisted surgery learning curve assessed through the reduction of procedure times | Through study completion, on average 1 year
  Assessment of the Robotic assisted surgery learning curve through an assessment of procedure times
Procedure times | Day of surgical intervention
  The duration of each procedure will be registered. Mean duration will be estimated
Intra- and post-operative complications | Day of surgical intervention, 24h post-surgery and after 30-day follow-up
  The number of intra- and post-operative complications complications will be registered and described
Post-operative pain | End of surgery to 24 hours post-op
  Post-operative pain will be reported by the patients through a 10-points VAS scale (1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Professor, Principal Investigator — Department for the Protection of Health of Women, Newborns, Children and Adolescents A. Gemelli University Polyclinic Catholic University of the Sacred Heart
Locations (1):
- Department for the Protection of Health of Women, Newborns, Children and Adolescents A. Gemelli University Polyclinic Catholic University of the Sacred Heart, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schreuder HW, Verheijen RH. Robotic surgery. BJOG. 2009 Jan;116(2):198-213. doi: 10.1111/j.1471-0528.2008.02038.x. PMID 19076952
- [Background] Murphy DG, Hall R, Tong R, Goel R, Costello AJ. Robotic technology in surgery: current status in 2008. ANZ J Surg. 2008 Dec;78(12):1076-81. doi: 10.1111/j.1445-2197.2008.04754.x. PMID 19087046
- [Background] Heemskerk J, van Gemert WG, de Vries J, Greve J, Bouvy ND. Learning curves of robot-assisted laparoscopic surgery compared with conventional laparoscopic surgery: an experimental study evaluating skill acquisition of robot-assisted laparoscopic tasks compared with conventional laparoscopic tasks in inexperienced users. Surg Laparosc Endosc Percutan Tech. 2007 Jun;17(3):171-4. doi: 10.1097/SLE.0b013e31805b8346. PMID 17581459
- [Background] Nezhat C, Saberi NS, Shahmohamady B, Nezhat F. Robotic-assisted laparoscopy in gynecological surgery. JSLS. 2006 Jul-Sep;10(3):317-20. PMID 17212887
- [Background] Advincula AP, Song A. The role of robotic surgery in gynecology. Curr Opin Obstet Gynecol. 2007 Aug;19(4):331-6. doi: 10.1097/GCO.0b013e328216f90b. PMID 17625414
- [Background] Marchal F, Rauch P, Verhaeghe JL, Guillemin F. [Laparoscopic surgery and robot]. Bull Cancer. 2007 Dec;94(12):1075-80. doi: 10.1684/bdc.2007.0524. French. PMID 18156116
- [Background] De Ugarte DA, Etzioni DA, Gracia C, Atkinson JB. Robotic surgery and resident training. Surg Endosc. 2003 Jun;17(6):960-3. doi: 10.1007/s00464-002-8745-6. Epub 2003 Mar 28. PMID 12658424
- [Background] Weinberg L, Rao S, Escobar PF. Robotic surgery in gynecology: an updated systematic review. Obstet Gynecol Int. 2011;2011:852061. doi: 10.1155/2011/852061. Epub 2011 Nov 28. PMID 22190948
- [Background] Ercoli A, D'asta M, Fagotti A, Fanfani F, Romano F, Baldazzi G, Salerno MG, Scambia G. Robotic treatment of colorectal endometriosis: technique, feasibility and short-term results. Hum Reprod. 2012 Mar;27(3):722-6. doi: 10.1093/humrep/der444. Epub 2012 Jan 11. PMID 22238113
- [Background] Carvalho L, Abrao MS, Deshpande A, Falcone T. Robotics as a new surgical minimally invasive approach to treatment of endometriosis: a systematic review. Int J Med Robot. 2012 Jun;8(2):160-5. doi: 10.1002/rcs.451. Epub 2011 Dec 9. PMID 22162096
- [Background] Yim GW, Kim YT. Robotic surgery in gynecologic cancer. Curr Opin Obstet Gynecol. 2012 Feb;24(1):14-23. doi: 10.1097/GCO.0b013e32834daebc. PMID 22123220
- [Background] Fagotti A, Gagliardi ML, Fanfani F, Salerno MG, Ercoli A, D'Asta M, Tortorella L, Turco LC, Escobar P, Scambia G. Perioperative outcomes of total laparoendoscopic single-site hysterectomy versus total robotic hysterectomy in endometrial cancer patients: a multicentre study. Gynecol Oncol. 2012 Jun;125(3):552-5. doi: 10.1016/j.ygyno.2012.02.035. Epub 2012 Mar 3. PMID 22391483